CLINICAL TRIAL: NCT00592202
Title: Laparoscopic Adjustable Gastric Banding as a Treatment for Morbid Obesity in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Bob Kanard, Visiting Assistant Professor/MD, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0732
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Morbid Obesity
Keywords: Morbid obesity; Adolescents; Gastric restrictive procedure; Adjustable gastric band; Treatment
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Adolescents between the ages 14 through 17 with a BMI of 40 or more or with a BMI of 35 or more and with an obesity related comorbidity will undergo placement of an adjustable gastric band
  Interventions: Device: Placement of an adjustable gastric band

INTERVENTIONS:
Device: Placement of an adjustable gastric band — Laparoscopic placement of an adjustable gastric band around the upper portion of the stomach and subsequent adjustments of the band via a subcutaneous port as needed to maintain appropriate restriction.

SUMMARY:
The purpose of this study is to determine whether the LAP-BAND system is safe and effective in morbidly obese adolescents.

DETAILED DESCRIPTION:
The aim of this research is to evaluate the safety and efficacy of the use of the Lap-Band system in the morbidly obese adolescent population in the United States. We also propose to take advantage of the opportunity for liver biopsy and the data collected for the FDA study in adolescents to answer several questions: 1) what is the true incidence of non-alcoholic fatty liver disease (NAFLD) and its variants in morbidly obese adolescents; 2) what is the course of the NAFLD disease in adolescents who have undergone weight loss, including the progression from steatosis to NASH/ fibrosis or the progression of NASH to cirrhosis? 3) What are the factors implicated in this progression and 4) Is there a link between the excess visceral fat, MS and NAFLD as assessed by parallel changes in metabolic syndrome (MS) and NAFLD following weight loss intervention. The LAPBAND may provide obese adolescents with a significantly less morbid and reversible surgical option for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Ages 14 through 17
* BMI greater than 40
* BMI 35 to 40 and also having an obesity related comorbidity
* Have a history of working in a multidisciplinary weight loss program utilizing nutritional training, behavior modification, and activity training

Exclusion Criteria:

* Subject history of congenital or acquired anomalies fo the gastrointestinal tract
* Severe cardiopulmonary or other serious organic disease
* Severe coagulopathy
* Hepatic insufficiency or cirrhosis
* History of bariatric gastric or esophageal surgery
* History of intestinal obstruction or adhesive peritonitis
* History of esophageal motility disorders
* Type I diabetes

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2004-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Weight loss | Every six months

SECONDARY OUTCOMES:
Resolution of comorbidities | every six months
Assess the status of comorbidities and changes in quality of life scores from baseline. | every six months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kanard, M.D., Principal Investigator — Division of Pediatric Surgery, UIC
Locations (1):
- UIMC, Chicago, Illinois, United States